CLINICAL TRIAL: NCT06214741
Title: A Phase III, Randomized, Double-blind, Parallel-group, Efficacy and Safety Study of BI 456906 Administered Subcutaneously Compared With Placebo in Chinese Participants With a BMI >=28 kg/m2 or BMI >=24 kg/m2 With at Least One Weight-related Complication
Brief Title: A Study to Test Whether Survodutide (BI 456906) Helps Chinese People Living With Overweight or Obesity to Lose Weight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404-0061; U1111-1295-9567 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- survodutide 3.6 mg (Experimental)
  Interventions: Drug: survodutide
- survodutide 4.8 mg (Experimental)
  Interventions: Drug: survodutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 456906

INTERVENTIONS:
Drug: survodutide — once weekly subcutaneous injection
  Other Names: BI 456906
  Arms: survodutide 3.6 mg; survodutide 4.8 mg
Drug: Placebo matching BI 456906 — Once weekly subcutaneous injection
  Arms: Placebo

SUMMARY:
This study in China is open to adults who are at least 18 years old who are living with overweight or obesity. People with a body mass index (BMI) of 28 kg/m^2 or higher or 24 kg/m^2 or higher with at least 1 weight related problem can join the study. The main purpose of this study is to find out whether a medicine called survodutide helps people with overweight or obesity. 2 different doses of survodutide are tested in this study.

Participants are put into 3 groups by chance. Each participant has an equal chance of being in each group. 2 groups get different doses of survodutide. 1 group gets placebo. Participants get survodutide or placebo as injections under the skin once a week for about 19 months.

Placebo injections look like survodutide injections but do not contain any medicine.

Participants are in the study for about 21 months. During this time, there are 20 visits. 14 visits are in person at the study site. Where possible, 6 visits can be done by video call, or by phone in rare cases. During this time, doctors regularly measure participant's body weight. Results are compared between the survodutide groups and placebo group to see whether the treatment works. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 years at the time of signing informed consent.
2. Body mass index (BMI) ≥28 kg/m^2 at screening, OR BMI ≥24 kg/m^2 at screening with the presence of at least one of the following weight-related complications:

   * Hypertension (defined as repeated, i.e. at least 3 measurements in resting condition, systolic blood pressure (SBP) values of ≥140 mmHg and/or diastolic blood pressure (DBP) values of ≥90 mmHg in the absence of anti-hypertensive treatment, or intake of at least 1 anti-hypertensive drug to maintain a normotensive blood pressure)
   * Dyslipidaemia (defined as at least 1 lipid-lowering treatment required to maintain normal blood lipid levels, or low density lipoprotein (LDL) cholesterol ≥160 mg/dL (≥4.1 mmol/L), or triglycerides ≥150 mg/dL (≥1.7 mmol/L), or high density lipoprotein (HDL) cholesterol <40 mg/dL (<1.0 mmol/L) for men or HDL cholesterol <50 mg/dL (<1.3 mmol/L) for women)
   * Obstructive sleep apnoea
   * Cardiovascular disease (CVD) (e.g. heart failure (HF) with New York Heart Association (NYHA) functional class II-III, history of ischaemic or haemorrhagic stroke or cerebrovascular revascularisation procedure [e.g. carotid endarterectomy and/or stent], myocardial infarction (MI), coronary artery disease, or peripheral vascular disease)
   * Type 2 diabetes mellitus (T2DM) diagnosed at least 180 days prior to screening (glycosylated haemoglobin A1c (HbA1c) ≥6.5% (48 mmol/mol) and <10% (86 mmol/mol), and fasting plasma glucose (FPG) ≤11.1 mmol/L measured by the central laboratory at screening

     --- Currently treated with either: diet and exercise alone or stable treatment (for at least 3 months prior to screening) with metformin, sodium-glucose cotransporter-2 inhibitor (SGLT2i) inhibitor, acarbose, sulfonylurea, or glitazone as single agent therapy, or up to 3 anti-hyperglycaemia medications (metformin, SGLT2i, acarbose, sulfonylurea, or glitazone) according to local label
   * Non-alcoholic steatohepatitis (NASH), as assessed in medical records by histological liver assessment (within the last 6 months)
3. History of at least one self-reported unsuccessful dietary effort to lose body weight
4. Signed and dated written informed consent in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
5. Woman of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria and instructions on the duration of their use will be provided in the participant information.

Further inclusion criteria apply.

Exclusion Criteria:

(A) Obesity:

1. Body weight change (self-reported) >5% within 3 months before screening.
2. Treatment with any medication for the indication obesity within 3 months before screening.
3. Previous or planned (during the trial period) treatment for obesity with surgery or a weight loss device, or prior surgery of the GI tract that could interfere with body weight The following are allowed: (1) liposuction and/or abdominoplasty, if performed >1 year before screening, (2) lap banding, if the band has been removed >1 year before screening, (3) intragastric balloon, if the balloon has been removed >1 year before screening, (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed >1 year before screening, (5) appendectomy, (6) simple hernia repair, or (7) cholecystectomy
4. Have obesity induced by other endocrinologic disorders (for example, Cushing Syndrome) or diagnosed monogenetic or syndromic forms of obesity (for example, melanocortin 4 receptor deficiency, leptin deficiency, or Prader Willi Syndrome) (B) Diabetes-related for participants with T2DM:
5. Treatment with any medication for the indication of T2DM other than stated in the inclusion criteria within 3 months before screening (i.e. insulin, amylin analogues, glucagon-like peptide-1 receptor (GLP- 1R)) agonists, GLP-1R agonist/insulin/glucose-dependent insulinotropic polypeptide (GIP) combinations, and dipeptidyl peptidase 4 inhibitor (DPP-4i))
6. New initiation of any other glucose-lowering investigational drug within 3 months prior to screening for this trial
7. Uncontrolled and potentially unstable diabetic retinopathy or maculopathy, verified by an eye examination within 3 months prior to screening or in the period between screening and randomisation Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline to Week 52 | At baseline and at Week 52.
Achievement of body weight reduction ≥5% (yes/no) from baseline to Week 52 | At baseline and at Week 52.

SECONDARY OUTCOMES:
Key secondary endpoint: Achievement of body weight reduction ≥10% (yes/no) from baseline to Week 52 | At baseline and at Week 52
Key secondary endpoint: Achievement of body weight reduction ≥15% (yes/no) from baseline to Week 52 | At baseline and at Week 52
Key secondary endpoint: Absolute change from baseline to Week 52 in waist circumference (cm) | At baseline and at Week 52
Achievement of body weight reduction ≥20% (yes/no) from baseline to Week 52 | At baseline and at Week 52
Absolute change from baseline to Week 52 in body weight (kg) | At baseline and at Week 52
Absolute change from baseline to Week 52 in glycosylated haemoglobin A1c (HbA1c) (%) | At baseline and at Week 52
Absolute change from baseline to Week 52 in HbA1c (mmol/mol) | At baseline and at Week 52
Absolute change from baseline to Week 52 in systolic blood pressure (SBP) (mmHg) | At baseline and at Week 52
Absolute change from baseline to Week 52 in diastolic blood pressure (DBP) (mmHg) | At baseline and at Week 52
Absolute change from baseline to Week 52 in body mass index (BMI) (kg/m^2) | At baseline and at Week 52
Absolute change from baseline to Week 52 in fasting plasma glucose (FPG) (mg/dL) | At baseline and at Week 52
Absolute change from baseline to Week 52 in fasting plasma insulin (FPI) (mIU/L) | At baseline and at Week 52
Absolute change from baseline to Week 52 in total cholesterol (mg/dL) | At baseline and at Week 52
Absolute change from baseline to Week 52 in high-density lipoprotein (HDL) cholesterol (mg/dL) | At baseline and at Week 52
Absolute change from baseline to Week 52 in low-density lipoprotein (LDL) cholesterol (mg/dL) | At baseline and at Week 52
Absolute change from baseline to Week 52 in very low-density lipoprotein (VDL) cholesterol (mg/dL) | At baseline and at Week 52
Absolute change from baseline to Week 52 in triglycerides (mg/dL) | At baseline and at Week 52
Absolute change from baseline to Week 52 in free fatty acids (mg/dL) | At baseline and at Week 52
Absolute change from baseline to Week 52 in alanine aminotransferase (ALT) (U/L) | At baseline and at Week 52
Absolute change from baseline to Week 52 in aspartate aminotransferase (AST) (U/L) | At baseline and at Week 52

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - Beijing Chao-Yang Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Pinggu Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Second Hospital of Jilin University, Changchun
  - Changzhou Second People's Hospital, Changzhou
  - People's Hospital of Sichuan Province, Chengdu
  - Second Affiliated Hospital Chongqing Medical University, Chongqing
  - NanFang Hosptial, Guangzhou
  - Forth Clinical Hospital of Harbin Medical University, Harbin
  - Huzhou Central Hospital, Huzhou
  - Center Hospital of Jinan, Jinan
  - Jincheng General Hospital, Jincheng
  - Lishui Municipal Central Hospital, Lishui
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Panjin Liao Oil Gem Flower Hospital, Panjin
  - Shanghai Fifth People's Hospital affiliated to Fudan University, Shanghai
  - Siping Central People's Hospital, Siping
  - Tianjin Medical University Chu Hisen-I Memorial Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an
  - The People's Hospital Of Xuancheng City, Xuancheng
  - Yichang Central People's Hospital, Yichang
  - Yueyang People's Hospital, Yueyang

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com